CLINICAL TRIAL: NCT05332717
Title: Association Between Melatonin Use and Improved Sleep Quality After Total Knee Arthroplasty: A Randomized Control Trial
Brief Title: TKA Melatonin and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-0150
Record Dates: First submitted 2021-08-10; First posted 2022-04-18 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Arthroplasty; Replacement; Knee; Sleep Initiation and Maintenance Disorders
Keywords: Melatonin; Arthroplasty; Knee; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: This study will compare postoperative sleep quality in two groups of patients undergoing primary total knee arthroplasty (TKA):
  * Group 1 will take melatonin during the 6 week postoperative period
  * Group 2 will take a placebo during the 6 week postoperative period
Who Masked: Participant
Masking Description: Participants will not be informed if they are receiving study drugs or placebo pills.
  Placebos will be compounded to be identical to treatment drugs in shape, size, color, texture etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin Group (Experimental) (Experimental): Patients who will take one (1) 5mg Melatonin tablet 30 minutes before bedtime daily for the 6 weeks following surgery.
  Interventions: Dietary Supplement: Melatonin 5 mg
- Placebo Group (Control) (Sham Comparator): Patients who will take one (1) placebo (Vitamin C) tablet 30 minutes before bedtime daily for the 6 weeks following surgery.
  Interventions: Dietary Supplement: Placebo (Vitamin C)

INTERVENTIONS:
Dietary Supplement: Melatonin 5 mg — Participants will be taking one 5 mg tablet of Melatonin 30 minutes before bedtime nightly, for 6 weeks following their knee replacement surgeries.
  Arms: Melatonin Group (Experimental)
Dietary Supplement: Placebo (Vitamin C) — Participants will be taking one placebo tablet 30 minutes before bedtime nightly, for 6 weeks following their knee replacement surgeries.
  Arms: Placebo Group (Control)

SUMMARY:
This randomized controlled trial (RCT) will compare the effects of melatonin vs. placebo in patients undergoing primary total knee arthroplasty (TKA). This RCT aims to study the effects melatonin has on sleep quality after TKA. Patients will be blinded to their respective groups and will be instructed to take either 5mg melatonin or a placebo pill (Vitamin C) for 6 weeks postoperative. Sleep quality surveys will be administered preoperatively and post-operative week 6, 90-days and 1 year. Poor sleep quality is a common issue faced by patients undergoing TKA. The goal of this study is see if melatonin can improve postoperative sleep quality, and if so, does improved sleep quality correlate to improvements in other postoperative outcomes.

DETAILED DESCRIPTION:
This study will compare postoperative sleep quality in two groups of patients undergoing primary total knee arthroplasty (TKA):

* Group 1 will take one melatonin (5 mg) tablet nightly, ~30 minutes before bedtime during the 6 week postoperative period
* Group 2 will take one placebo (5 mg Vitamin C) tablet nightly, ~30 minutes before bedtime during the 6 week postoperative period

The primary outcome will be sleep quality at 6 weeks. Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI). The survey will be administered preoperatively, 6-weeks, 90-days and 1 year postoperatively. Preoperative surveys will be completed in-person, on-site by study participants. All postoperative surveys will be distributed via email.

Secondary outcomes include:

* (KOOS Jr, LEAS, VR-12, VAS) administered preoperatively, at 6-weeks, 90-days and 1-year post-operatively.
* Total opioids prescribed in first 3 months postoperative will be collected using iStop
* Frequency of CMS defined surgicalcomplications in the first 90-days after primary TKA.
* Adverse events of Melatonin during the first 6 weeks (collected via email survey sent to participants once per week, for the first 6 weeks)
* Study medication compliance at 6 weeks (collected via email survey sent to participants once per week, for the first 6 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary, unilateral TKA
* Primary diagnosis of osteoarthritis (OA)
* Aged 18+
* Subject is opioid naive (has not taken opioids during the 6 months prior to surgery)
* Subject is not currently taking sleep medication
* English speaking
* Has working email (for survey purposes)

Exclusion Criteria:

* Patients with diagnosis other than OA including: Inflammatory arthritis; Post-traumatic OA; Chronic pain; Insomnia*; Depression*; Anxiety*; Any active sleep disorder
* Planned contralateral knee or subsequent total joint arthroplasty within 90 days
* Any planned surgery within 90 days
* Patient taking medication for depression or insomnia or anxiety during the 6 months prior to surgery
* Patients with renal or hepatic disorders as these can affect melatonin metabolism

  * Insomnia, anxiety, and depression will be defined as use of controlled medication for that disorder which will be identified in istop or HSS record of the patient filled in the 6 months prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | Preoperatively
  Assessed based on self-reported data collected using the Pittsburgh Sleep Quality Index (PSQI). Minimum Score: 0; Maximum Score: 21. Higher scores indicate a worse outcome.
Sleep Quality | 6-week
  Assessed based on self-reported data collected using the Pittsburgh Sleep Quality Index (PSQI). Minimum Score: 0; Maximum Score: 21. Higher scores indicate a worse outcome.
Sleep Quality | 90 days
  Assessed based on self-reported data collected using the Pittsburgh Sleep Quality Index (PSQI). Minimum Score: 0; Maximum Score: 21. Higher scores indicate a worse outcome.
Sleep Quality | 1-year
  Assessed based on self-reported data collected using the Pittsburgh Sleep Quality Index (PSQI). Minimum Score: 0; Maximum Score: 21. Higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Knee Function | Preoperatively, 6-week, 90-day and 1-year follow-up
  Assessed based on self-reported data collected using the abbreviated Knee Injury and Osteoarthritis Outcome Score (KOOS Jr). Minimum Score: 0; Maximum Score: 28. Higher scores indicate a better outcome.
Lower Extremity Activity | Preoperatively, 6-week, 90-day and 1-year follow-up
  Assessed based on self-reported data collected using the Lower Extremity Activity Scale (LEAS). Minimum Score: 1; Maximum Score: 18. Higher scores indicate a better outcome.
Overall Health | Preoperatively, 6-week, 90-day and 1-year follow-up
  Assessed based on self-reported data collected using the Veterans Rand 12 (VR-12) Scale. Minimum Score: 0; Maximum Score: 100. Higher scores indicate a better outcome.
Pain Ratings | Preoperatively, 6-week, 90-day and 1-year follow-up
  Assessed based on self-reported data collected using the Visual Analogue Pain Scale. Minimum Score: 0; Maximum Score: 10. Higher scores indicate a worse outcome.
Opioids Prescribed | 90-day follow-up
  This will me quantified in morphine milligram equivalents (MMEs). This information will be obtained for each patient using institutionally queried i-Stop data.
Quantity of Postoperative Centers for Medicare and Medicaid Services Complications | 90-day follow-up
  Assessed using institutional medical record data.
Study Medication Compliance | Weekly (Up to 6 weeks)
  Assessed based on self-reported data collected via study survey.
Quantity of Adverse Melatonin Medical Events | Weekly (Up to 6 weeks)
  Assessed based on self-reported data collected via study survey.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro G Della Valle, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available at the study conclusion due to its inclusion of Protected Healthcare Information (PHI).

REFERENCES:
- [Background] Shakya H, Wang D, Zhou K, Luo ZY, Dahal S, Zhou ZK. Prospective randomized controlled study on improving sleep quality and impact of zolpidem after total hip arthroplasty. J Orthop Surg Res. 2019 Sep 3;14(1):289. doi: 10.1186/s13018-019-1327-2. PMID 31481074
- [Background] Mammoto T, Fujie K, Taguchi N, Ma E, Shimizu T, Hashimoto K. Short-Term Effects of Early Postoperative Celecoxib Administration for Pain, Sleep Quality, and Range of Motion After Total Knee Arthroplasty: A Randomized Controlled Trial. J Arthroplasty. 2021 Feb;36(2):526-531. doi: 10.1016/j.arth.2020.08.018. Epub 2020 Aug 18. PMID 32900564
- [Background] Kirksey MA, Yoo D, Danninger T, Stundner O, Ma Y, Memtsoudis SG. Impact of Melatonin on Sleep and Pain After Total Knee Arthroplasty Under Regional Anesthesia With Sedation: A Double-Blind, Randomized, Placebo-Controlled Pilot Study. J Arthroplasty. 2015 Dec;30(12):2370-5. doi: 10.1016/j.arth.2015.06.034. Epub 2015 Jun 21. PMID 26173613
- [Background] Luo ZY, Li LL, Wang D, Wang HY, Pei FX, Zhou ZK. Preoperative sleep quality affects postoperative pain and function after total joint arthroplasty: a prospective cohort study. J Orthop Surg Res. 2019 Nov 21;14(1):378. doi: 10.1186/s13018-019-1446-9. PMID 31752947
- [Background] Hemati K, Pourhanifeh MH, Dehdashtian E, Fatemi I, Mehrzadi S, Reiter RJ, Hosseinzadeh A. Melatonin and morphine: potential beneficial effects of co-use. Fundam Clin Pharmacol. 2021 Feb;35(1):25-39. doi: 10.1111/fcp.12566. Epub 2020 Jun 21. PMID 32415694
- [Background] Oh ES, Leoutsakos JM, Rosenberg PB, Pletnikova AM, Khanuja HS, Sterling RS, Oni JK, Sieber FE, Fedarko NS, Akhlaghi N, Neufeld KJ. Effects of Ramelteon on the Prevention of Postoperative Delirium in Older Patients Undergoing Orthopedic Surgery: The RECOVER Randomized Controlled Trial. Am J Geriatr Psychiatry. 2021 Jan;29(1):90-100. doi: 10.1016/j.jagp.2020.05.006. Epub 2020 May 16. PMID 32532654

DOCUMENTS (1):
  • Informed Consent Form (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT05332717/ICF_000.pdf